CLINICAL TRIAL: NCT01124539
Title: A Phase 2 Study of AR-67 (7-t-butyldimethylsiltyl-10-hydroxy-camptothecin) in Adult Patients With Recurrence of Glioblastoma Multiforme (GBM) or Gliosarcoma
Brief Title: Study of AR-67 in Adult Patients With Recurrence of Glioblastoma Multiforme (GBM) or Gliosarcoma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Arno Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ARN-AR67-IIS202
Record Dates: First submitted 2010-05-12; First posted 2010-05-17 (Estimated); Last update posted 2014-12-09 (Estimated); Status verified 2014-01

CONDITIONS: Glioblastoma Multiforme; GBM; Gliosarcoma
Keywords: Adult Patients; Recurrence of Glioblastoma Multiforme; Recurrence of GBM; Gliosarcoma
MeSH Terms: conditions — Glioblastoma; Gliosarcoma | interventions — 7-tert-butyldimethylsilyl-10-hydroxycamptothecin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- AR-67 (Experimental)
  Interventions: Drug: AR-67 (7-t-butyldimethylsiltyl-10-hydroxy-camptothecin)

INTERVENTIONS:
Drug: AR-67 (7-t-butyldimethylsiltyl-10-hydroxy-camptothecin) — IV AR-67 administered once daily for 5 days on an every 21-day cycle
  Other Names: AR67; formerly DB-67; formerly DB67

SUMMARY:
The primary objective of this study is to determine the 6-month Progression free survival (PFS) when intravenous (IV) AR-67 is administered in adults with confirmed recurrence of GBM who have not recently (> 90 days) recurred after treatment bevacizumab (including patients who've received temazolamide, but no bevacizumab). The primary objective in the rapid bevacizumab failure group (< 90 days) is to determine the 2-month PFS.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female age 18 years or older.
2. Patient, or legal representative, able to provide study-specific informed consent after risks and benefits of treatment have been explained prior to screening.
3. Confined histopathology of World Health Organization (WHO) Grade IV GBM or Gliosarcoma at primary diagnosis or recurrence by local pathology review.
4. Unequivocal radiographic evidence of recurrence of tumor by MRI within 14 days prior to enrollment.
5. Patients who have progressed, had surgery, and have no measurable disease are eligible as long as they have adequately recovered from the surgery.
6. Received prior radiotherapy and temozolomide treatment.
7. Received last chemotherapy or biologic therapy treatment ≥14 days before first dose of study drug (≥42 days if nitrosourea or ≥90 days if bevacizumab for the non-bevacizumab failure cohort or therapeutic antibody was administered) or, for daily type regimens, ≥7 days or 5 half-lives of the drugs' pharmacokinetics/dynamics or biologic activities, whichever is longer, before the first dose of study drug. For subjects that have received prior chemotherapy, all toxicities need to have resolved ≤ Grade 1 prior to the administration of study drug. For the patients in the bevacizumab failure cohort, failure must have occurred within the prior 90 days of receiving the last bevacizumab dose.
8. Completed radiotherapy ≥90 days before study starts.
9. Completed the administration of any investigational agent ≥14 days or 5 half-lives of the drugs' PK/dynamics or biologic activities, whichever is longer, before study starts.
10. Karnofsky performance status of ≥60%.
11. Recovered to Grade 1 or less from the toxic effects of any earlier intervention.
12. Patients receiving EIADs must be switched to non-EIADs at least 14 days prior to study start.
13. Adequate renal, liver, and bone marrow function according to the following criteria:

    * Absolute neutrophil count ≥1500/mcL
    * Platelets ≥150,000/mcL
    * Total bilirubin within upper limit of normal (ULN)
    * Aspartate aminotransferase (AST) ≤ 2.5 X institutional ULN
    * Creatinine within normal limits or creatinine clearance ≥ 50 mL/min for patients with creatinine levels above normal limits.
14. Demonstrated, in the opinion of the investigator, the ability to follow directions necessary to participate in the clinical trial.
15. Women of childbearing potential must agree to use acceptable contraceptive methods as follows:

    * An intrauterine device with a documented failure rate of less than 1% per year.
    * Vasectomized partner who is sterile prior to the female patient's entry and is the sole sexual partner for that female.
    * Complete abstinence from sexual intercourse for 14 days before exposure to investigational product, through the dosing period, and for at least 21 days after the last dose of investigational product.
    * Double-barrier contraception (condom with spermicidal jelly, foam suppository, or film; diaphragm with spermicide, or male condom and diaphragm with spermicide).

    Note: These methods are to be used consistently and in accordance with both the product label and the instructions of the treating physician. Oral contraceptives are not reliable due to potential drug-drug interactions and should be used with caution if the patient insists on their use as a contraceptive.
16. A life expectancy of greater than 2 months.

Exclusion Criteria:

1. Patients on therapeutic Coumadin; however, patients on therapeutic Coumadin that can switch to low molecular weight heparin (LMWH) at least 7 days prior to first dosing will be eligible for study participation.
2. Female patients who are pregnant or breastfeeding.
3. Prior malignancy other than curatively treated basal cell or cervical carcinoma in situ or adequately treated Stage I or II cancer from which the patient is currently in complete remission and from which the patient has been disease-free for three years.
4. Uncontrolled concurrent illness including active infection requiring intravenous antibiotics, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
5. Known HIV infection.
6. Any other condition that would compromise treatment and/or evaluation with reasonable safety.
7. Completed intracranial surgery ≤ 14 days before the study starts.
8. Received an anti-epilpetic drug, which is a CYP3A4 inducer from ≤ 14 days prior to screening until study end. See Appendix 1 for the list of enzyme inducing anti-epileptic drugs.

   Inducers of CYP3A4 may also alter the metabolism of AR-67. The following list of CYP3A4 inducers are prohibited from 14 days prior to screening through discontinuation from the study:
   * HIV: efavirenz, nevirapine
   * Antibiotics: rifampin (rifampicin), rifabutin, rifapentine
   * Antiretrovirals: efavirenz, nevirapine
   * Miscellaneous: St. John's Wort, modafinil
   * Anti-Epileptic Drugs: phenytoin, phenobarbital, primidone, carbamazapine, oxcarbazapine and topiramate
9. Co-administration of AR-67 and medications that are substrates for the CYP450 enzymes and have the potential to cause serious and/or life-threatening AE's is prohibited. These medications include (but are not limited to):

   * Anticoagulants: therapeutic coumadin
   * Oral hypoglycemics: glilpizide, glyburide, tolbutamide, glimepiride, nateglinice
   * Erectile dysfunction agents: sildenafil, tadalafil, vardenafil
   * Ergot derivatives: dihydroergotamine, ergonovine, ergotamine, methylergonovine
   * Neuroleptics: pimozide
   * Antiarrhythmics: bepridil, flecainide, lidocaine, meziletine, amiodarone, quinidine, propafenone
   * Immune modulators: cyclosporine, tacrolimus, sirolimus
   * Miscellaneous: theophylline, quetiapine, risperidone, tacrine, clozapine, atomoxetine
10. The following list of CYP3A4 inhibitors are prohibited from 14 days prior to screening through discontinuation from the study:

    * Antibiotics: clarithromycin, erythromycin, troleandomycin
    * HIV: antiretrovirals (delaviridine), protease inhibitors (ritonavir, indinavir, saquinavir, nelfinavir, amprenavir, lopinavir)
    * Antifungals: itraconazole, ketoconazole, voriconazole, fluconazole (>150 mg daily)
    * Antidepressants: nefazodone, fluvoxamine
    * Calcium channel blockers: verapamil, diltiazem
    * Gastrointestinal: cimetidine, aprepitant
    * Miscellaneous: grapefruit or its juice
11. Progressive disease with any topoisomerase I inhibitors.
12. History of anaphylactic injection reaction of > Grade 3 to any product used to formulate AR-67.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Estimated)
Dates: Start 2009-12; Primary Completion 2014-09 (Actual); Study Completion 2015-02 (Estimated)

PRIMARY OUTCOMES:
Determine the 6-month Progression free survival (PFS) AR-67 is administered in adults with confirmed recurrence of GBM who have not recently (> 90 days) recurred after treatment bevacizumab. | 6 month PFS
  Thirty-two (32) patients will be accrued to the non-bevacizumab failure cohort.
The primary objective in the rapid bevacizumab failure group (< 90 days) is to determine the 2-month PFS. | 2 month PFS
  26 subjects will be enrolled in the second cohort (Rapid Avastin Progressors).

SECONDARY OUTCOMES:
the effect of AR-67 on overall survival (OS) | 1 year
the effect of AR-67 on overall PFS | 6 Months
the effect of AR-67 on event-free survival (EFS) | 6 Months
the impact of AR-67 on tumor response in patients with measurable disease | 6 Months
the safety and tolerability of AR-67 | 6 Months

CONTACTS AND LOCATIONS:
Overall Officials: James J Vredneburgh, MD, Principal Investigator — Duke University Medical Center - The Preston Robert Tisch Brain Tumor Center
Locations (9):
- United States (7):
  - Northwestern University - Robert H Lurie Comprehensive Cancer Center, Chicago, Illinois
  - University of Kentucky - Markey Cancer Center, Lexington, Kentucky
  - North Shore - Long Island Jewish Hospital/Monter Cancer Center, Lake Success, New York
  - Duke University Medical Center - The Preston Robert Tisch Brain Tumor Center, Durham, North Carolina
  - Derrick L Davis Forsyth Regional Cancer Center, Winston-Salem, North Carolina
  - The Ohio State University - James Comprehensive Cancer Center, Columbus, Ohio
  - University of Utah - Huntsman Cancer Center, Salt Lake City, Utah
- Canada (2):
  - University of Calgary - Tom Baker Cancer Center, Calgary, Alberta
  - University of Alberta - Cross Cancer Institute, Edmonton, Alberta